CLINICAL TRIAL: NCT00055185
Title: Safety and Efficacy of PRO 542 in the Treatment of HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT2001; 5R44AI048278-05 (NIH)
Record Dates: First submitted 2003-02-20; First posted 2003-02-21 (Estimated); Last update posted 2008-10-03 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infections; Acquired Immune Deficiency Syndrome
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — CD4-IgG(2)

INTERVENTIONS:
Drug: CD4-IgG2 (PRO 542)

SUMMARY:
The purpose of this study is to determine any adverse effects of PRO 542 after administration and to determine the anti-HIV effects of PRO 542 in the patient.

DETAILED DESCRIPTION:
A 2 arm study involving a series of 3 triweekly doses of PRO 542. One arm will involve patients on a stable dose of anti-retroviral therapy and the other arm will consist of patients not receiving anti-retroviral therapy. Three patients will be enrolled in each arm followed by a safety evaluation. Following the safety evaluation, 3 more patients may be enrolled in each arm. After the first 12 patients, an additional 12 patients may be enrolled pending safety data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HIV
* Patients must be on a stable dose of acceptable anti-HIV therapy or receiving no anti-HIV therapy for at least four (4) weeks prior to the start of this study
* HIV-1 determination by RNA-PCR greater than or equal to 100,000 copies/ml
* CD4 count >50/cubic mm at screening

Exclusion Criteria:

* Patients who have previously received PRO 542
* Patients with active, significant infection (other than HIV) not controlled by antibiotics
* Pregnant or lactating women
* Patients with an estimated life expectancy of <3 months
* Patients currently receiving steroids or other immunosuppressive therapy or immunoglobulin therapy except for topical or inhaled steroids
* Patients with known allergy or hypersensitivity to PRO 542 or immunoglobulin preparations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-04; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery M Jocbson, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States